CLINICAL TRIAL: NCT06839456
Title: Phase 1/2 Study: CD45RA Depleted Peripheral Stem Cell Addback to Prevent Viral and Fungal Infections Following Alternative Donor TCRab/CD19 Depleted Hematopoietic Stem Cell Transplant
Brief Title: Phase 1/2: CD45RA Depleted Stem Cell Addback to Prevent Viral or Fungal Infections Post TCRab/CD19 Depleted HSCT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Timothy Olson, Medical Director, Hematopoietic Stem Cell Transplantation (HSCT) Program, Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-022264
Record Dates: First submitted 2025-02-16; First posted 2025-02-21 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Leukemia; High Risk Acute Lymphoblastic Leukemia; High Risk Acute Myeloid Leukemia; Relapse Leukemia; MDS (Myelodysplastic Syndrome); Relapsed Non-Hodgkin Lymphoma; Acquired Aplastic Anemia; Inherited BMF Syndrome; Immunodeficiency; Primary Immune Regulatory Disorder; Hemoglobinopathies; Bone Marrow Failure; Inborn Errors of Metabolism; HLH
Keywords: alpha beta T cell depletion; CD45RA; CD45RO; GVHD prevention; Memory T cells
MeSH Terms: conditions — Leukemia; Anemia, Refractory, with Excess of Blasts; Lymphoma, Non-Hodgkin; Congenital Bone Marrow Failure Syndromes; Immunologic Deficiency Syndromes; Hemoglobinopathies; Bone Marrow Failure Disorders; Metabolism, Inborn Errors | interventions — Clinical Trials, Phase I as Topic

STUDY DESIGN:
Intervention Model Description: Use of CliniMACS based system for TCRαβ/CD19 Depleted Peripheral Stem Cells and CD45RA Depleted Peripheral Stem Cell Addback.
  Approximately 90% of the peripheral stem cell (PSC) product will be processed using the CliniMACS system for TCRαβ and CD19 cell depletion. In addition, approximately 10% of the PSCs will undergo CD45RA depletion also using the CliniMACS system. Processing is completed in accordance with the Investigator Brochure and Technical Manual following the laboratory standard operating procedures (SOPs) and using aseptic technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Phase 1:TCRab/CD19 depleted PSCT with CD45RA depleted addback using mismatched related donors (MMRD) (Experimental): Stem cell source: mobilized peripheral blood stem cells (PBSC)
  Donor type: > or = 5/10 mismatched related donor
  Conditioning: disease specific standard of care (SOC) regimens
  Interventions: Device: Phase 1 Dose Level 1; Device: Phase 1 Dose Level 2; Device: Phase 1 Dose Level 3
- Phase 2:TCRab/CD19 depleted PSCT with CD45RA depleted addback at MTD found in phase 1 using MMRD (Experimental): Stem cell source: mobilized PBSC
  Donor type: > or = 5/10 mismatched related donor
  Conditioning: disease specific SOC regimens
  Interventions: Device: Phase 2 Maximum Tolerated Dose determined in Phase 1
- Phase 2:TCRab/CD19 depleted PSCT with CD45RA depleted addback using unrelated donors (Experimental): Stem cell source: mobilized PBSC
  Donor type: 9/10 or 10/10 matched unrelated donor
  Conditioning: disease specific SOC regimens
  Interventions: Device: Phase 2 Established Dose from prior study, NCT03810196

INTERVENTIONS:
Device: Phase 1 Dose Level 1 — Patients in the first dose level for the CD45RA depleted addback will receive 1 X 10^6 CD45RO+ T cells/kg. Once all patients in this dose group have been evaluated for acute GVHD at day 100, then we will advance to the next dose level if indicated by safety analysis.
  Arms: Phase 1:TCRab/CD19 depleted PSCT with CD45RA depleted addback using mismatched related donors (MMRD)
Device: Phase 1 Dose Level 2 — Patients in the second dose level for the CD45RA depleted addback will receive 2 X 10^6 CD45RO+ T cells/kg. Once all patients in this dose group have been evaluated for acute GVHD at day 100, then we will advance to the next dose level if indicated by safety analysis.
  Arms: Phase 1:TCRab/CD19 depleted PSCT with CD45RA depleted addback using mismatched related donors (MMRD)
Device: Phase 1 Dose Level 3 — Patients in the third and final dose level for the CD45RA depleted addback will receive 5 X 10^6 CD45RO+ T cells/kg. All patients in this dose group will be evaluated for acute GVHD at day 100. Based on these findings, the maximum tolerated dose (MTD) will be determined.
  Once MTD for the addback cell dose has been determined in Phase 1, subjects with mismatched related donors will then enroll in Phase 2.
  Arms: Phase 1:TCRab/CD19 depleted PSCT with CD45RA depleted addback using mismatched related donors (MMRD)
Device: Phase 2 Maximum Tolerated Dose determined in Phase 1 — Patients with mismatched related donors will receive the CD45RA depleted addback at the maximum tolerated dose determined in the Phase 1 portion of the study.
  Arms: Phase 2:TCRab/CD19 depleted PSCT with CD45RA depleted addback at MTD found in phase 1 using MMRD
Device: Phase 2 Established Dose from prior study, NCT03810196 — Patients with unrelated donors will receive the CD45RA depleted addback at the dose 5 X 10^6 CD45RO+ T cells.
  Arms: Phase 2:TCRab/CD19 depleted PSCT with CD45RA depleted addback using unrelated donors

SUMMARY:
The major morbidities of allogeneic hematopoietic stem cell transplant (HSCT) using donors that are not human leukocyte antigen (HLA) matched siblings are graft vs host disease (GVHD) and life- threatening infections. T cell receptor alpha beta (TCRαβ) T lymphocyte depletion and CD19+ B lymphocyte depletion of alternative donor hematopoietic stem cell (HSC) grafts is effective in preventing GVHD, but immune reconstitution may be delayed, increasing the risk of infections. The central hypothesis of this study is that an addback of CD45RO memory T lymphocytes, derived from a fraction of the original donor peripheral stem cell product depleted of CD45RA naïve T lymphocytes, will accelerate immune reconstitution and help decrease the risk of infections in TCRab/CD19 depleted PSCT.

DETAILED DESCRIPTION:
The risk of severe graft versus host disease (GVHD) is increased with the use of unrelated and partially matched related donors. T cell depletion reduces the risk of severe GVHD, but immune reconstitution is delayed. Important memory T cells that may protect patients from fungal and viral infections are also removed in the T depletion process. CD45RA depletion has been studied both as a single step to reduce the risk of GVHD, and also, in conjunction with αβTCR depleted hematopoietic stem cell grafts to accelerate immune reconstitution. This single institutional trial builds on data from our protocol #18-015286, NCT03810196, "CD45RA Depleted Peripheral Stem Cell Addback for Patients at Risk for Viral or Fungal Infections Post-TCRαβ/CD19 Depleted Hematopoietic Stem Cell Transplant". This prior protocol was limited to patients with hematologic malignancies using only unrelated donors as the stem cell source.

This new study will broaden the eligible diagnoses to include non-malignant transplant indications and participants with greater than or equal to 5/10 HLA matched related donors (also known as haploidentical).

This will be a phase 1 and phase 2 study depending on the donor type. Phase 1 will include patients receiving cells from mismatched/haploidentical related donors. This will be a dose escalation study to determine the maximum tolerated cell dose of the CD45RA depleted addback. Once that dose is determined, patients with this donor type will be treated as part of phase 2.

Patients receiving their cells from unrelated donors ( 9/10 or 10/10 HLA matched) will be treated as part of phase 2 with the CD45RA depleted addback cell dose that was used on our prior study. Phase 1 and phase 2 will run concurrently.

ELIGIBILITY:
Inclusion Criteria:

1. Disease for which allogeneic HSCT may be curative.
2. Remission status of hematologic malignancies and additional disease-specific eligibility determinations will be according to standards of practice within the CHOP Cellular Immunotherapy and Transplant Program (CTTS).
3. Patients must be 25 years of age and less
4. Evaluation for organ and infectious status as per our CTTS standard operating procedure.
5. Signed consent by parent/guardian or able to give consent if 18 years of age and older.
6. Participants of childbearing potential must have a negative pregnancy test as per institutional SOP.

Exclusion Criteria:

1. Patients who have performance score less than 60.
2. No suitable donor available for mobilized peripheral stem cells.
3. Patients with Hodgkin lymphoma or non-Burkitt, non-lymphoblastic lymphoma.
4. Planned receipt of alemtuzumab during conditioning.
5. Patients with an available 10/10 HLA matched sibling donor.
6. Patients who do not meet institutional disease, organ or infectious criteria.

Donor selection and eligibility:

1. Unrelated donor meets National Marrow Donor Program criteria for donation.
2. Related donor (at least haploidentical) willing and able to donate mobilized peripheral stem cells.
3. HLA testing/matching

   * HLA testing to be done by molecular methods for A, B, C, DRB1, DQB1
   * Related donor: Must be ≥ 5/10 match
   * Unrelated donor: 10/10 or 9/10 match
   * KIR typing for haploidentical donor for hematologic malignancies
   * Donor specific HLA antibodies (DSA) should be assessed for all subjects receiving an HLA mismatched graft (≤ 9/10).
4. Donor must be willing to undergo granulocyte colony stimulating factor (GCSF) mobilization and peripheral blood stem cell collection
5. Donors must be willing to sign consent to participate in this study.

Ages: 1 Month to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate number of patients with acute graft vs host disease (aGVHD) | Up to 100 days post-transplantation
  Safety evaluation assessment by cumulative incidence of acute graft vs host disease (reaction of donor immune cells against host tissues) to determine percentage of patients that develop grade 3-4 aGVHD.
Evaluate number of patients with chronic graft vs host disease (cGVHD) | Up to 2 years post-transplantation
  Safety evaluation assessment by cumulative incidence and severity of chronic GVHD (graft vs host disease that occurs more than 100 days after transplant) to determine percentage of patients that develop cGVHD.

SECONDARY OUTCOMES:
Evaluate time to immune reconstitution | 2 years
  Evaluate time to achievement of standard immune reconstitution benchmarks following TCRαβ/CD19 depleted HSCT with CD45RA+ depleted addback, compared to historical experience with TCRαβ/CD19 depletion alone.
Evaluate number of patients with viral reactivation | 2 years
  Evaluate number of patients with viral reactivation (CMV, adenovirus, EBV, BK) following TCRαβ/CD19 depleted HSCT with CD45RA depleted addback, compared to historical experience with TCRαβ/CD19 depletion alone.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Olson, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No